CLINICAL TRIAL: NCT00347919
Title: A Phase II, Open-Label, Randomized, Multicenter Trial of GW786034 (Pazopanib) in Combination With Lapatinib (GW572016) Compared to Lapatinib Alone as First Line Therapy in Subjects With Advanced or Metastatic Breast Cancer With ErbB2 Fluorescence In Situ Hybridization (FISH) Positive Tumors
Brief Title: Pazopanib Plus Lapatinib Compared To Lapatinib Alone In Subjects With Advanced Or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VEG20007
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Results first posted 2011-02-21 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-01

CONDITIONS: Neoplasms, Breast
Keywords: GW786034; Quality of Life; GW572016; Lapatinib; Pazopanib; Metastatic; Breast cancer; Genetics; FISH; Advanced
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — pazopanib; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- monotherapy arm (Experimental): 1500 mg (6 x 250 mg tablets) oral lapatinib once daily
  Interventions: Drug: lapatinib (GW572016) 1500 mg
- Cohort 1 combination arm (Experimental): 1000 mg (4 x 250 mg tablets) of oral lapatinib and 400 mg (4 x 100 mg tablets) of oral pazopanib taken together once daily
  Interventions: Drug: pazopanib (GW786034) 400 mg; Drug: lapatinib (GW572016) 1000 mg
- Cohort 2 combination arm (Experimental): 1500 mg (6 x 250 mg tablets) of oral lapatinib and 800 mg (1 x 500 mg tablets plus 3 x 100 mg tablets) of oral pazopanib taken together once daily
  Interventions: Drug: lapatinib (GW572016) 1500 mg; Drug: pazopanib (GW786034) 800 mg

INTERVENTIONS:
Drug: pazopanib (GW786034) 400 mg — 400 mg administered orally once daily
  Arms: Cohort 1 combination arm
Drug: lapatinib (GW572016) 1500 mg — 1500 mg administered orally once daily.
  Arms: Cohort 2 combination arm; monotherapy arm
Drug: lapatinib (GW572016) 1000 mg — 1000 mg administered orally once daily
  Arms: Cohort 1 combination arm
Drug: pazopanib (GW786034) 800 mg — 800 mg administered orally once daily
  Arms: Cohort 2 combination arm

SUMMARY:
This study is being conducted to compare the efficacy and safety of pazopanib in combination with lapatinib with that of lapatinib alone in subjects with locally advanced or metastatic breast cancer whose tumors overexpress the ErbB2 protein.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria apply:
* Women ≥ 18 years of age with a life expectancy of ≥ 12 weeks.
* Note: National Institute of Neurological and Communicative Disorders and Stroke (NINCDS) and Alzheimer's Disease and Related Disorders Association (ADRDA).)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
* Histologically confirmed invasive breast cancer with incurable stage IIIb, stage IIIc with T4 lesion, or stage IV disease at primary diagnosis or at relapse after curative-intent surgery.
* No prior chemotherapy, immunotherapy, biologic therapy or anti-ErbB1/ErbB2 therapy for metastatic or recurrent disease (other than neoadjuvant or adjuvant therapy). Prior hormonal therapy (e.g., tamoxifen, raloxifen or an aromatase inhibitor) for advanced or metastatic disease is permitted provided at least 2 weeks have elapsed between the completion of the prior therapy and start of study drugs.
* Note: Subjects must have documented progressive disease (PD) or be intolerant to hormonal therapy. This must be documented in the source documentation.
* Prior neoadjuvant therapy and/or adjuvant therapy is permitted.
* Note:
* (a) Subjects who have received both neoadjuvant and adjuvant therapies must have at least 6 months between completion of the chemotherapy-component of adjuvant therapy and start of study drug(s)
* (b) Subjects who have received only adjuvant therapy must have at least 6 months between completion of the chemotherapy-component of adjuvant therapy and start of study drug(s)
* (c) Subjects who have received only neoadjuvant therapy must have at least 6 months between completion of neoadjuvant therapy and start of study drug(s)
* (d) Subjects who have received trastuzumab or hormonal agents as all or part of adjuvant therapy are eligible provided: (1) 2 weeks have elapsed since last dose (2) 6 months have elapsed between the start of trastuzumab or hormonal therapy and start of study drugs.
* Radiotherapy prior to initiation of randomized therapy to a limited area (e.g., palliative treatment for painful disease) other than the sole site of measurable and assessable disease is allowed however, subjects must have completed treatment at least 4 weeks prior to starting study drugs, and must have recovered from all treatment-related toxicities prior to starting pazopanib and/or lapatinib.
* Documented amplification of ErbB2 by Fluorescence In Situ Hybridization (FISH) in either the primary or metastatic tumor tissue. Archived tumor tissue must be provided for ErbB2 FISH testing by the central laboratory, which will be used to determine eligibility.
* Note: Subjects that have documented ErbB2 amplification based on prior FISH testing or documented ErbB2 overexpression based on prior immunohistochemistry (IHC) with a value of 3+ are eligible, however, archived tumor tissue must be provided for confirmation by the central laboratory. If the results from prior testing are not confirmed by the central laboratory, then the subject can continue to receive study drug(s) at the discretion of the investigator, but will be excluded from the statistical analysis.
* Archived tumor tissue (paraffin-embedded) must be available to correlate tumor response with intra-tumoral genetic changes as well as expression levels of relevant biomarkers. Results of biomarkers will not be used to determine subject eligibility for the study.
* Ability to swallow and retain oral medication.
* Disease must be measurable according to Response Evaluation Criteria in Solid Tumors (RECIST).
* Subjects must have chosen treatment with lapatinib and/or pazopanib as initial treatment over other initial treatments (such as cytotoxic chemotherapy regimens or trastuzumab as a single agent) for locally advanced or metastatic disease.
* Adequate organ function as defined below:
* System (Laboratory Values)
* Hematologic:Absolute neutrophil count (ANC) (≥1.5 X 109/L) Platelets (≥100 X 109/L)
* Hepatic:Albumin(≥2.5 g/dL)Serum bilirubin(≤1.5 X upper limit of normal (ULN) unless due to Gilbert's syndrome) aspartate aminotransferase (AST) and alanine aminotransferase (ALT) (≤2.0 X ULN)
* Renal:Calculated creatinine clearance1 (≥50 mL/min) Urine Protein2
* (Negative, trace or +1 by dipstick urinalysis or <1.0 gram determined by 24 hour urine protein analysis).
* A patient should first be screened with dipstick urinalysis. If urine protein by dipstick analysis is≥2+, then a 24-hour urine protein must be assessed and 24 hour urine protein must be <1 g protein to be eligible.
* Cardiac ejection fraction within the institutional range of normal as measured by echocardiogram. Multigated acquisition (MUGA) scans will be accepted in cases where an echocardiogram cannot be performed or is inconclusive or where MUGA scans are the accepted standard. Subjects with known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure are not eligible.
* A female is eligible to enter and participate in this study if she is of:
* Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had:
* A hysterectomy
* A bilateral oophorectomy (ovariectomy)
* A bilateral tubal ligation
* Is post-menopausal (total cessation of menses for ≥1 year)
* Childbearing potential, has a negative serum pregnancy test within 2 weeks of the first dose of study medication, and agrees to use adequate contraception during study participation and for a minimum of 2 menstrual cycles after the last dose of study medication. GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows:
* An intrauterine device with a documented failure rate of less than 1% per year.
* Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
* Complete abstinence from sexual intercourse for 14 days before exposure to investigation product, through the clinical trial, and for at least 2 menstrual cycles after the last dose of investigational product.
* Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide).
* Oral contraceptives are not reliable due to the potential drug-drug interactions.
* Subjects must complete all screening assessments as outlined in the protocol.
* Subjects must provide written informed consent prior to performance of any study-specific procedures or assessments and are willing to comply with treatment and follow-up.

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Subjects with bilateral breast cancer or bone metastases as the only disease site.
* Patients with high disease burden defined as >30% replacement of hepatic parenchyma with metastases, symptomatic pulmonary metastases (e.g., clinically significant dyspnea, cough, or chest pain attributable to pulmonary metastases), or >3 visceral organs with tumor involvement.
* History of other malignancy. Subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Sarcoma histology.
* Concurrent disease or condition that would make the subject inappropriate for study participation including (1) any unresolved or unstable, serious toxicity from prior administration of another investigational drug, (2) any serious medical disorder that would interfere with the subject's safety, obtaining informed consent or compliance to the study.
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously treated CNS metastases, are asymptomatic, and have had no requirement for steroids or antiseizure medication for ³ 2 months prior to study enrollment. Routine screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases.
* Malabsorption Syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel.
* Active peptic ulcer disease, inflammatory bowel disease, or other gastrointestinal condition increasing the risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 4 weeks prior to beginning therapy.
* Presence of uncontrolled infection.
* Concurrent cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, hormonal therapy, and tumor embolization).
* Concurrent treatment with an investigational agent or participation in another clinical trial.
* Use of an investigational anti-cancer drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of pazopanib and/or lapatinib.
* Prior use of an investigational or licensed drug that targets either vascular endothelial growth factor (VEGF) or VEGF receptors, or ErbB2 (except for trastuzumab when used in the neo-adjuvant/adjuvant setting).
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib or lapatinib.
* Has taken/is taking prohibited medications, Lapatinib-related, orPazopanib-related.
* Corrected QT interval (QTc) prolongation defined as QTc interval > 480 msecs.
* History of any one of the following cardiac conditions within the past 6 months:
* Cardiac angioplasty or stenting
* Myocardial infarction
* Unstable angina
* History of cerebrovascular accident within the past 6 months.
* Poorly controlled hypertension (systolic blood pressure (SBP) of ≥140mmHg, or diastolic blood pressure (DBP) of ≥90mmHg).
* Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. The blood pressure (BP) must be re-assessed on two occasions that are separated by a minimum of 24 hours. The mean SBP/DBP values from both BP assessments must be < 140/90mmHg in order for a subject to be eligible for the study.
* Presence of any non-healing wound, fracture, or ulcer, or the presence of symptomatic peripheral vascular disease.
* Evidence of bleeding diathesis or coagulopathy.
* Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks prior to beginning therapy, or anticipation of the need for a major surgical procedure during the course of the study; minor surgical procedures such as fine needle aspiration or core biopsy within 1 week prior to beginning therapy are also excluded.
* Pregnant or lactating female.
* Has Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* History of untreated deep venous thrombosis (DVT) within the past 6 months (e.g. calf vein thrombosis).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2006-07; Primary Completion 2008-08 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (75):
- United States (19):
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Alhambra, California
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Oxnard, California
  - GSK Investigational Site, Redondo Beach, California
  - GSK Investigational Site, Santa Barbara, California
  - GSK Investigational Site, Santa Maria, California
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Lubbock, Texas
  - GSK Investigational Site, San Antonio, Texas
- Canada (3):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Weston, Ontario
- France (7):
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Hyères
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille Cedex BP 156
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Strasbourg
- Hungary (2):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Győr
- India (6):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Delhi
  - GSK Investigational Site, Jaipur
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Trivandrum
- Israel (6):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Rehovot
  - GSK Investigational Site, Tel Aviv
- Malaysia (2):
  - GSK Investigational Site, Bandar Tun Razak, Cheras
  - GSK Investigational Site, Petaling Jaya
- Mexico (2):
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, Mexico City
- Pakistan (4):
  - GSK Investigational Site, Islamabad
  - GSK Investigational Site, Karachi
  - GSK Investigational Site, Lahore
  - GSK Investigational Site, Multan
- Peru (2):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, Callao
- Poland (5):
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Warsaw
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- GSK Investigational Site, Singapore, Singapore
- South Korea (4):
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seodaemun-gu, Seoul
  - GSK Investigational Site, Songpa-gu, Seoul
  - GSK Investigational Site, Suwon, Kyonggi-do
- GSK Investigational Site, Bangkok, Thailand
- United Kingdom (9):
  - GSK Investigational Site, Chelmsford, Essex
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Sutton, Surrey
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Ipswich
  - GSK Investigational Site, London
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Plymouth

REFERENCES:
- [Background] Johnston SR, Gomez H, Stemmer SM, Richie M, Durante M, Pandite L, Goodman V, Slamon D. A randomized and open-label trial evaluating the addition of pazopanib to lapatinib as first-line therapy in patients with HER2-positive advanced breast cancer. Breast Cancer Res Treat. 2013 Feb;137(3):755-66. doi: 10.1007/s10549-012-2399-4. Epub 2013 Jan 3. PMID 23283526
- [Derived] de Jonge MJ, Hamberg P, Verweij J, Savage S, Suttle AB, Hodge J, Arumugham T, Pandite LN, Hurwitz HI. Phase I and pharmacokinetic study of pazopanib and lapatinib combination therapy in patients with advanced solid tumors. Invest New Drugs. 2013 Jun;31(3):751-9. doi: 10.1007/s10637-012-9885-8. Epub 2012 Oct 6. PMID 23054212

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) were enrolled into two cohorts. Cohort 1: Par. were randomized 1:1 to lapatinib 1500 mg or lapatinib 1000 mg/pazopanib 400 mg. Cohort 2: After enrollment was complete for Cohort 1, par. were enrolled to lapatinib 1500 mg/pazopanib 800 mg. All par. who received study drug are accounted for in the Participant Flow module.
Pre-assignment Details: Female par. with >=18 years of age with histologically confirmed invasive breast cancer were enrolled in the study. Total 189 par. (Cohort 1, combination n = 76, lapatinib n = 73; Cohort 2, n = 40) received study drug.
Groups:
- Cohort 1: Lapatinib 1500 mg: Lapatinib 1500 milligrams (mg) administered orally once a day
- Cohort 1: Lapatinib 1000 mg/Pazopanib 400 mg: Lapatinib 1000 mg and Pazopanib 400 mg administered orally once a day
- Cohort 2: Lapatinib 1500 mg/Pazopanib 800 mg: Lapatinib 1500 mg and Pazopanib 800 mg administered orally once a day
Period: Overall Study
Arm/Group | Cohort 1: Lapatinib 1500 mg | Cohort 1: Lapatinib 1000 mg/Pazopanib 400 mg | Cohort 2: Lapatinib 1500 mg/Pazopanib 800 mg
Started | 73 (Safety Population) | 76 (Safety Population) | 40 (Safety Population)
Completed | 2 | 0 | 2
Not Completed | 71 | 76 | 38
Not completed — Lost to Follow-up | 11 | 13 | 0
Not completed — Withdrawal by Subject | 6 | 8 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Sponsor terminated study | 15 | 10 | 16
Not completed — Death | 35 | 42 | 19
Not completed — Par. Started Other Treatment | 1 | 1 | 1
Not completed — Missing | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Lapatinib 1500 mg | Cohort 1: Lapatinib 1000 mg/Pazopanib 400 mg | Cohort 2: Lapatinib 1500 mg/Pazopanib 800 mg | Total
Number analyzed (Participants) | 72 | 69 | 36 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] — The data in the Participant Flow module are for the Safety Population, comprised of any participant who had received study drug. All of the Baseline data are from a more limited population: the Modified Intent-to-Treat Population (MITT), comprised of those participants who received study drug and who also were confirmed to be Human Epidermal growth factor Receptor 2 (ErbB2) positive by fluorescent in situ hybridization (FISH) analysis.
  years | 53.5 (11.20) | 52.1 (12.76) | 54.1 (12.93) | 52.8 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants] — Males were excluded. All participants were female.
  Participants
    Female | 72 | 69 | 36 | 177
    Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 0 | 1 | 0 | 1
  American Indian or Alaska Native | 20 | 18 | 0 | 38
  Asian | 33 | 30 | 3 | 66
  White | 19 | 18 | 32 | 69
  Other | 0 | 1 | 0 | 1
  Unknown | 0 | 1 | 1 | 2
Child-Bearing Potential [Number; unit: participants]
  Post-Menopausal | 49 | 46 | 22 | 117
  Sterile (of child-bearing age) | 3 | 2 | 5 | 10
  Potentially able to bear children | 20 | 21 | 9 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progressive Disease at Week 12 in Cohort 1
Description: The percentage of participants with progressive disease (PD) 12 weeks after randomization was measured. Per Response Evaluation Criteria In Solid Tumors (RECIST), a response of PD is defined as a >=20% increase in target lesions. Participants were also classified as having PD if their response at Week 12 was unknown or missing. Response was determined by an independent radiologist and by an investigator.
Time Frame: Week 12
Population: Cohort 1: Modified Intent-to-Treat (ITT) Population (all randomized, centrally confirmed, ErbB2 FISH-positive participants).
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Lapatinib 1500 mg | Cohort 1: Lapatinib 1000 mg/Pazopanib 400 mg
Number analyzed (Participants) | 72 | 69
percentage of participants
  Independently Evaluated | 38.9 | 36.2
  Investigator Evaluated | 43.1 | 37.7
Statistical Analysis 1: Comparison: Cohort 1: Lapatinib 1500 mg vs Cohort 1: Lapatinib 1000 mg/Pazopanib 400 mg; Test type: Superiority or Other; p = 0.3724, Chi-squared; Percentage difference = 2.7, 90% CI [-11.0 to 16.3] — Difference in the percentage of independently-evaluated PD between lapatinib and combination therapy (lapatinib plus pazopanib)
Statistical Analysis 2: Comparison: Cohort 1: Lapatinib 1500 mg vs Cohort 1: Lapatinib 1000 mg/Pazopanib 400 mg; Test type: Superiority or Other; p = 0.2578, Chi-squared; Percentage difference = 5.4, 90% CI [-8.4 to 19.2] — Difference in the percentage of investigator-evaluated PD between lapatinib and combination therapy (lapatinib plus pazopanib)

2. Secondary Outcome: Overall Survival for Cohort 1
Description: Overall survival (OS) is defined as the time from randomization until death due to any cause. Participants who are alive as of the date of last contact are censored. There was insufficient follow-up to adequately assess OS for Cohort 2. Median OS cannot be presented for the lapatinib arm because the upper bound of the 95% confidence interval is undefined due to insufficient follow-up.
Time Frame: Randomization until death due to any cause (up to 106.43 weeks)
Population: MITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 1: Lapatinib 1500 mg | Cohort 1: Lapatinib 1000 mg/Pazopanib 400 mg | Cohort 2: Lapatinib 1500 mg/Pazopanib 800 mg
Number analyzed (Participants) | 0 | 69 | 0
weeks |  | 91.0 [69.4 to 91.0] |
Statistical Analysis 1: Comparison: Cohort 1: Lapatinib 1500 mg vs Cohort 1: Lapatinib 1000 mg/Pazopanib 400 mg; Test type: Superiority or Other; p = 0.7488, Log Rank

3. Secondary Outcome: Response at Week 12 for Cohort 1 and Cohort 2
Description: The percentage of participants achieving either a complete (CR) or partial (PR) tumor response per Response Evaluation Criteria in Solid Tumors (RECIST) is presented. CR, all detectable tumor has disappeared; PR, a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum; Progressive disease (PD), a >=20% increase in target lesions; Stable Disease, small changes that do not meet previously given criteria. IRC, independent review committee. Participants with an unknown or missing response were treated as non-responders.
Time Frame: Week 12
Population: MITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Lapatinib 1500 mg | Cohort 1: Lapatinib 1000 mg/Pazopanib 400 mg | Cohort 2: Lapatinib 1500 mg/Pazopanib 800 mg
Number analyzed (Participants) | 72 | 69 | 36
percentage of participants
  Complete response, IRC evaluated | 0 | 0 | 0
  Complete response, Investigator evaluated | 1 | 0 | 0
  Partial response, IRC evaluated | 22 | 36 | 33
  Partial response, Investigator evaluated | 26 | 45 | 50
  Stable disease, IRC evaluated | 39 | 28 | 31
  Stable disease, Investigator evaluated | 29 | 17 | 14
  Progressive disease, IRC evaluated | 17 | 20 | 8
  Progressive disease, Investigator evaluated | 38 | 20 | 11
  Unknown/missing, IRC evaluated | 22 | 15 | 28
  Unknown/missing, Investigator | 6 | 17 | 25

4. Secondary Outcome: Duration of Response in Cohort 1
Description: Duration of response is defined as the length of time from the time from the first observation of response until progression of disease or death. Duration of response depends on two things: (1) when response is counted as starting; (2) when response is counted as ending.There were insufficient data to adequately assess duration of response for Cohort 2. IRC, independent review committee. For participants who do not progress or die, duration of response was censored at the date of last adequate assessment.
Time Frame: Time from first documented evidence of complete or partial response until the first documented sign of disease progression or death due to any cause (up to 106.71 weeks)
Population: MITT Population
Measure: Median (Inter-Quartile Range); unit: weeks
Groups:
- Cohort 2: Lapatinib 1500 mg/ Pazopanib 800 mg: Lapatinib 1500 mg and Pazopanib 800 mg administered orally once a day
Arm/Group | Cohort 1: Lapatinib 1500 mg | Cohort 1: Lapatinib 1000 mg/Pazopanib 400 mg | Cohort 2: Lapatinib 1500 mg/ Pazopanib 800 mg
Number analyzed (Participants) | 72 | 69 | 0
weeks | 27.1 [24.3 to 27.7] | 24.3 [12.3 to 24.3] |

5. Secondary Outcome: Time to Response (Complete or Partial Response) in Cohort 1 and Cohort 2
Description: Time to response is defined as the time from randomization to the time of first documented evidence of a complete (CR) or partial response (PR). The time to response will depend on when the response is counted as starting. Per RECIST: CR, all detectable tumor has disappeared; PR, a >=30% decrease in the sum of the target dimensions of the target lesions taking as a reference the baseline sum.
Time Frame: The time from randomization to the time of first documented evidence of complete or partial response (up to 81.14 weeks for Cohort 1 and 44.29 weeks for Cohort 2)
Population: MITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 1: Lapatinib 1500 mg | Cohort 1: Lapatinib 1000 mg/Pazopanib 400 mg | Cohort 2: Lapatinib 1500 mg/Pazopanib 800 mg
Number analyzed (Participants) | 72 | 69 | 36
weeks
  IRC Evaluated | 8.1 [7.9 to 11.4] | 8.3 [8.0 to 11.9] | 8.3 [7.4 to 8.7]
  Investigator Evaluated | 8.0 [7.9 to 8.1] | 8.1 [8.0 to 8.4] | 8.0 [7.3 to 8.6]

6. Secondary Outcome: Percentage of Participants With Progressive Disease at Week 12
Description: The percentage of participants with progressive disease (PD) 12 weeks after randomization was measured. Participants were classified as having PD if their response at Week 12 was unknown or missing. Per Response Evaluation Criteria In Solid Tumors (RECIST), PD is defined as a >=20% increase in target lesions. IRC, independent review committee.
Time Frame: Week 12
Population: Cohort 2 MITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 2: Lapatinib 1500 mg/Pazopanib 800 mg
Number analyzed (Participants) | 36
percentage of participants
  PD+Missing+Unknown, IRC evaluated | 36
  PD+Missing+Unknown, Investigator Evaluated | 36

ADVERSE EVENTS:
Time Frame: Study Entry until 28 days after the last dose.
Arm/Group | Cohort 1: Lapatinib 1500 mg | Cohort 1: Lapatinib 1000 mg/Pazopanib 400 mg | Cohort 2: Lapatinib 1500 mg/Pazopanib 800 mg
Serious Adverse Events (participants affected / at risk) | 10/73 | 18/76 | 13/40
Other Adverse Events (participants affected / at risk) | 63/73 | 71/76 | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Lapatinib 1500 mg (N=73) | Cohort 1: Lapatinib 1000 mg/Pazopanib 400 mg (N=76) | Cohort 2: Lapatinib 1500 mg/Pazopanib 800 mg (N=40)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 4 (4)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 3 (3) | 2 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Lapatinib 1500 mg (N=73) | Cohort 1: Lapatinib 1000 mg/Pazopanib 400 mg (N=76) | Cohort 2: Lapatinib 1500 mg/Pazopanib 800 mg (N=40)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 4 (10) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 6 (8) | 2 (10)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 2 (3)
Hypothyroidism (Endocrine disorders) | 0 (0) | 6 (7) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 8 (8) | 3 (3) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 7 (7) | 11 (14)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 7 (7) | 3 (4)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 41 (81) | 52 (172) | 34 (86)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 6 (9) | 8 (10) | 7 (8)
Nausea (Gastrointestinal disorders) | 13 (18) | 23 (31) | 28 (35)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 5 (6) | 5 (22) | 5 (7)
Vomiting (Gastrointestinal disorders) | 6 (10) | 15 (28) | 13 (19)
Asthenia (General disorders) | 9 (13) | 9 (11) | 5 (5)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 3 (3)
Chest pain (General disorders) | 0 (0) | 0 (0) | 4 (4)
Fatigue (General disorders) | 7 (7) | 12 (18) | 23 (25)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (10) | 6 (7) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (7)
Urinary tract infection (Infections and infestations) | 7 (8) | 4 (6) | 2 (2)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 3 (4)
Alanine aminotransferase increased (Investigations) | 13 (21) | 25 (39) | 15 (20)
Aspartate aminotransferase increased (Investigations) | 13 (16) | 26 (40) | 15 (22)
Blood bilirubin increased (Investigations) | 3 (4) | 10 (17) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 7 (8)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 3 (6)
Crystal urine present (Investigations) | 0 (0) | 5 (5) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 4 (5) | 0 (0)
Weight decreased (Investigations) | 3 (4) | 8 (10) | 5 (6)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 10 (10) | 9 (9) | 5 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 4 (11) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (5)
Decreased appetite (Metabolism and nutrition disorders) | 10 (12) | 17 (21) | 14 (21)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (8) | 4 (4) | 5 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9) | 9 (13) | 4 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 6 (6) | 4 (5) | 7 (10)
Dysgeusia (Nervous system disorders) | 1 (1) | 12 (13) | 12 (12)
Headache (Nervous system disorders) | 7 (12) | 6 (14) | 11 (15)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 8 (10) | 5 (5)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (2) | 8 (12) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (8) | 2 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (9) | 7 (10) | 13 (15)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 11 (13) | 10 (11)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (4) | 5 (5) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7) | 5 (5) | 2 (2)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 14 (14) | 11 (13)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (12) | 5 (5) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 21 (30) | 21 (27) | 16 (26)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Hypertension (Vascular disorders) | 4 (7) | 20 (25) | 15 (25)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 2 (3)

LIMITATIONS AND CAVEATS:
In 2008 at primary completion, study was terminated. In 2011, protocol amendment 4 (Am4), allowed continuation of treatment until PD for the 1 par. This par. completed the study per Am 4. Par. last visit occurred, the study is considered completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.